CLINICAL TRIAL: NCT02411149
Title: Adductor Canal Block and Functional Recovery After Total Knee Arthroplasty. A Double-Blind, Randomized Controlled Trial
Brief Title: Adductor Canal Block and Recovery After Total Knee Replacement Surgery
Acronym: ACB in TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-7016-A
Record Dates: First submitted 2015-03-30; First posted 2015-04-08 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Total Knee Arthroplasty
Keywords: Adductor Canal Block; Total Knee Arthroplasty
MeSH Terms: interventions — Ropivacaine; Epinephrine; Morphine; Anesthesia, Local; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Local Inflitration Only (Placebo Comparator): This group will receive LIA and saline solution (placebo) in the adductor canal block with NO morphine in the spinal anesthesia:
  * 30 ml normal saline
  * 3ml 0.5% preservative-free bupivacaine
  Interventions: Drug: Local Infiltration
- Adductor Canal Block (Active Comparator): This group will receive LIA and the standard local anesthetic in the ACB with NO morphine in the spinal anesthetic:
  * ropivacaine 0.5% with 1:400,000 epinephrine
  * 3ml 0.5% preservative-free bupivacaine
  Interventions: Drug: Adductor Canal Block
- Adductor Canal Block with Morphine (Active Comparator): This group will receive LIA with local anesthetic in the ACB and morphine in the spinal anesthetic:
  * ropivacaine 0.5% with 1:400,000 epinephrine
  * 3ml 0.5% preservative-free bupivacaine with 100mcg of intrathecal morphine (0.1ml of intrathecal morphine 1mg/ml)
  Interventions: Drug: Adductor Canal Block with Morphine

INTERVENTIONS:
Drug: Adductor Canal Block — Use of ropivacaine 0.5% with 1:400,000 epinephrine in the adductor canal along with a spinal anesthesia of 3ml 0.5% preservative-free bupivacaine.
  Other Names: ropivacaine with epinephrine
  Arms: Adductor Canal Block
Drug: Adductor Canal Block with Morphine — Use of ropivacaine 0.5% with 1:400,000 epinephrine in the adductor canal along with a spinal anesthesia of 3ml 0.5% preservative-free bupivacaine and 100mcg of intrathecal morphine (0.1ml of intrathecal morphine 1mg/ml)
  Other Names: ropivacaine with epinephrine and spinal intrathecal morphine
  Arms: Adductor Canal Block with Morphine
Drug: Local Infiltration — 30 ml normal saline in the adductor canal along with a spinal anesthesia of 3ml 0.5% preservative-free bupivacaine, in addition to the local infiltration.
  Other Names: saline
  Arms: Local Inflitration Only

SUMMARY:
This study aims to compare the functional recovery of patients undergoing Total Knee Arthroplasty based on the administration of an adductor canal block during their anesthesia treatment

DETAILED DESCRIPTION:
The period after total knee replacement (TKR) surgery is known to be painful for the first 24 hours, lasting up to 3 days in many cases. Successful management of pain after TKR is regarded as necessary to early recovery, rehabilitation and timely discharge. Severe pain following major joint arthroplasty can hinder early rehabilitation, may result in prolonged hospitalization and is a strong predictor of persistent pain beyond 3 months. Adequate analgesia following TKR is paramount to early recovery, rehabilitation and timely discharge. Therefore early postoperative analgesic and rehabilitation goals are intricately related.

Until now, different methods of pain treatment have been used, including intravenous narcotic pain medication, continuous femoral nerve block (numbing medication to a nerve in the thigh) and epidural analgesia (identical to the numbing method for childbirth). These are all effective methods but each is limited by side effects. In recent years, research has focused on administering local anesthetic further down in the leg, trying to minimize quadriceps muscle weakness while giving adequate pain relief after surgery. Local Infiltration Analgesia (LIA) and Adductor Canal Block (ACB) are examples of new farther sites of administration.

The purpose of this study is to determine which combination of analgesic interventions is the most effective treatment for pain and improvement in functional outcome for TKR.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status I-III
* 18 - 80 years of age
* BMI 18 - 40
* Scheduled for elective total knee replacement under spinal anesthesia
* Able to ambulate independently with a standard wheeled walker as maximum mobility aid

Exclusion Criteria:

* Revision knee arthroplasty
* Bilateral knee arthroplasty
* Lack of mental ability to provide informed consent
* Neuropathic pain or sensory disorders of the surgical limb
* Contraindication to regional anesthesia (intolerance to the study drugs, bleeding diathesis, coagulopathy, malignancy or infection at the site of block)
* Chronic opioid use defined as > 30 mg of daily oral morphine equivalents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test | 2-3 days post srugery
  TUG test reflects the time it takes a subject to stand up from a standard height armchair, walk 3 meters, walk back to the chair and sit down. It intends to assess a patient's global mobility as well as balance and risk of falling.

SECONDARY OUTCOMES:
Pain outcome - NRS | 2-3 days post surgery
  a) Pain scores assessed with an 11 point verbal numeric rating scale (NRS) where 0 is "no pain" and 10 is "the worst pain imaginable", both at rest and during active physiotherapy (measured daily for 3 days post-operatively) .
Analgesic outcomes - Cumulative systemic opioid consumption | 2-3 days post surgery
  Cumulative systemic opioid consumption measured as oral morphine mg equivalents (daily for 3 days post-operatively).
Analgesic outcomes - Proportion of patients who required "rescue" intravenous patient controlled analgesia | 2-3 days post surgery
  Proportion of patients who required "rescue" intravenous patient controlled analgesia (iv PCA) anytime in the post-operative period.
Analgesic outcomes - Incidence of opioid-related side effects | 2-3 days post surgery
  Incidence of opioid-related side effects
Secondary short-term physical and performance-based functional outcome measures - Proportion of patients achieving knee flexion range of motion (ROM) of 90 degrees | 2-3 days post surgery
  Proportion of patients achieving knee flexion range of motion (ROM) of 90 degrees (measured daily for 3 days post-operatively)
Secondary short-term physical and performance-based functional outcome measures - Distance walked | 2-3 days post surgery
  Distance walked
Secondary short-term physical and performance-based functional outcome measures - Hospital length of stay | 2-3 days post surgery
  Hospital length of stay
Secondary short-term physical and performance-based functional outcome measures - Discharge destination | 2-3 days post surgery
  Discharge destination (home or rehabilitation facility)
Medium-term self-reported functional outcome measures - WOMAC | baseline and 2-3 days post surgery
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) measured at baseline and at 3 months post-operatively
Medium-term self-reported functional outcome measures - LEFS | baseline and 2-3 days post surgery
  Lower extremity functional scale (LEFS) measured at baseline and at 3 months post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University of Toronto. University Health Network. Toronto Western Hospital.
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Puolakka PA, Rorarius MG, Roviola M, Puolakka TJ, Nordhausen K, Lindgren L. Persistent pain following knee arthroplasty. Eur J Anaesthesiol. 2010 May;27(5):455-60. doi: 10.1097/EJA.0b013e328335b31c. PMID 20299989
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Derived] Biswas A, Perlas A, Ghosh M, Chin K, Niazi A, Pandher B, Chan V. Relative Contributions of Adductor Canal Block and Intrathecal Morphine to Analgesia and Functional Recovery After Total Knee Arthroplasty: A Randomized Controlled Trial. Reg Anesth Pain Med. 2018 Feb;43(2):154-160. doi: 10.1097/AAP.0000000000000724. PMID 29315129